CLINICAL TRIAL: NCT01755468
Title: A Randomized Controlled Trial to Evaluate Early Intermittent Intensive Insulin Therapy as an Effective Treatment of Type 2 Diabetes: REmission Studies Evaluating Type 2 DM - Intermittent Insulin Therapy (RESET-IT Pilot Study)
Brief Title: Early Intermittent Intensive Insulin Therapy as an Effective Treatment of Type 2 Diabetes (RESET-IT Pilot Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-0263-A Pilot
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes
Keywords: beta-cell function, type 2 diabetes, intermittent insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous metformin (Active Comparator): After a 3-week course of intensive insulin therapy, participants will be treated with ongoing metformin monotherapy. Metformin will be initiated at 500mg twice a day for the first 2 weeks, before progressing to 1000mg twice a day for the duration of the trial (24 months).
  Interventions: Drug: Continuous metformin
- Intermittent insulin therapy (Experimental): After a 3-week course of intensive insulin therapy, participants will receive intermittent intensive insulin therapy for 2 weeks every 3 months. The 2-week course of insulin therapy will be repeated at 3-, 6-, 9-, 12-, 15-,18- and 21-months, with final outcome measurement performed at 24-months
  Interventions: Drug: Intermittent insulin therapy

INTERVENTIONS:
Drug: Intermittent insulin therapy
  Other Names: Basal insulin glargine and pre-meal insulin lispro
  Arms: Intermittent insulin therapy
Drug: Continuous metformin
  Other Names: Metformin
  Arms: Continuous metformin

SUMMARY:
Type 2 diabetes mellitus is a chronic metabolic disorder characterized by progressive deterioration in the function of the pancreatic beta-cells, which are the cells that produce and secrete insulin (the hormone primarily responsible for the handling of glucose in the body). The investigators propose a pilot randomized controlled trial to determine whether intermittent intensive insulin therapy is an effective therapeutic strategy that can preserve pancreatic beta-cell function and maintain glycemic control early in the course of type 2 diabetes.

DETAILED DESCRIPTION:
In this study, eligible patients with type 2 diabetes will be randomized to either intermittent insulin therapy or continuous metformin therapy, after both arms have first undergone a short course of intensive insulin therapy. The hypothesis under study is whether intermittent insulin therapy can better preserve beta-cell function.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 30 and 80 years inclusive
2. T2DM diagnosed by a physician </= 5 years prior to enrolment
3. Negative for anti-glutamic acid decarboxylase (anti-GAD) antibodies
4. On either no anti-diabetic medication or on metformin monotherapy, with no change in dose/regimen within 4 weeks prior to enrolment
5. A1c at screening between 5.5% and 9.0% inclusive if on metformin, or between 6.0% and 9.5% inclusive if on no oral anti-diabetic medication
6. BMI >/= 23 kg/m2
7. Negative pregnancy test at recruitment for all women with childbearing potential

Exclusion Criteria:

1. Current anti-diabetic treatment with insulin, sulfonylurea, thiazolidinedione, alpha-glucosidase inhibitor, GLP-1 agonist or dipeptidyl peptidase-4 inhibitor
2. Type 1 diabetes or secondary forms of diabetes
3. History of hypoglycemia unawareness or severe hypoglycemia requiring assistance
4. Any major illness with a life expectancy of <5 years
5. Hypersensitivity to insulin, metformin or the formulations of these products
6. Renal dysfunction as evidenced by estimated glomerular filtration rate (eGFR) <50 ml/min
7. Hepatic disease considered to be clinically significant (includes jaundice, chronic hepatitis, previous liver transplant) or transaminases >2.5 X upper limit of normal
8. History of congestive heart failure
9. Excessive alcohol consumption, defined as >14 alcoholic drinks per week for males and >9 alcoholic drinks per week for females
10. Unwillingness to administer insulin therapy or perform capillary blood glucose monitoring at least 4 times per day while receiving IIT
11. Pregnancy or unwillingness to use reliable contraception. Women should not be planning pregnancy for the duration of the study or the first 3 months after the study. Reliable contraception includes birth control pill, intra-uterine device, abstinence, tubal ligation, partner vasectomy, or condoms with spermicide.
12. Non-adherence to the induction phase or any factor likely to limit adherence to the study protocol, in the opinion of the investigator

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-04; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Baseline-adjusted beta-cell function at 2 years, measured by Insulin Secretion-Sensitivity Index-2 (ISSI-2). | 2 years
  ISSI-2 is an established measure of beta-cell function. ISSI-2 is defined as the product of (i) insulin secretion measured by the ratio of the area-under-the-insulin-curve to the area-under-the-glucose curve and (ii) insulin sensitivity measured by the Matsuda index.

SECONDARY OUTCOMES:
Baseline-adjusted glycemic control at 2-years. | 2 years
  The secondary outcome of baseline-adjusted glycemic control at 2-years will be assessed by A1c (glycated hemoglobin)

OTHER OUTCOMES:
Achievement of target glycemic control | 2 years
  Achievement of target glycemic control will be assessed by the proportion of participants with A1c <7.0%
achievement of glucose tolerance in the non-diabetic range | 2 years
  The proportion of participants with glucose tolerance in the non-diabetic range will be determined on oral glucose tolerance test (OGTT) and defined based on current Canadian Diabetes Association classifications for glucose tolerance status on OGTT.
achievement of normal glucose tolerance | 2 years
  The proportion of participants with normal glucose tolerance will be determined on oral glucose tolerance test (OGTT) and defined based on current Canadian Diabetes Association classifications for glucose tolerance status on OGTT.
insulin sensitivity | 2 years
  Insulin sensitivity will be measured by Matsuda index, a clamp-validated measure of whole-body insulin sensitivity that can be obtained from the oral glucose tolerance test

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Retnakaran, MD, Principal Investigator — Mount Sinai Hospital, Canada; Bernard Zinman, MD, Principal Investigator — Mount Sinai Hospital, Canada
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Retnakaran R, Choi H, Ye C, Kramer CK, Zinman B. Two-year trial of intermittent insulin therapy vs metformin for the preservation of beta-cell function after initial short-term intensive insulin induction in early type 2 diabetes. Diabetes Obes Metab. 2018 Jun;20(6):1399-1407. doi: 10.1111/dom.13236. Epub 2018 Feb 23. PMID 29377408